CLINICAL TRIAL: NCT00887848
Title: Effectiveness of Robotic Assisted Gait Training in Children With Cerebral Palsy: A Randomized Controlled Clinical Trial Including 3D Gait Analysis
Brief Title: Effectiveness of Robotic Assisted Gait Training in Children With Cerebral Palsy
Acronym: PeLoGAIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Reha Rheinfelden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PeLoGAIT_2009
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Palsy
Keywords: Child; Robotic-assisted treadmill training; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lokomat training (Experimental): Lokomat training
  Interventions: Other: Lokomat training
- Waiting list (Other): Lokomat training after waiting phase of 5 weeks
  Interventions: Other: Lokomat training

INTERVENTIONS:
Other: Lokomat training — 15 sessions of Lokomat training within 5 weeks (3 trainings/week)

SUMMARY:
The purpose of the study is to investigate the effectiveness of robotic-assisted locomotor therapy on improvements of functional gait parameters in ambulatory children with cerebral palsy.

DETAILED DESCRIPTION:
Within a randomized controlled design the effects of robotic-assisted locomotor training (15 sessions within 5 weeks) will be examined in a sample of 34 children with cerebral palsy.

Children will be randomly assigned to an intervention or waiting list group. Assessments will be performed at baseline, in week 6 as well as in week 12. The intervention is provided to the waiting list group after the assessment in week 6.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral spastic cerebral palsy
* Gross Motor Function Classification Scale (GMFCS) II-IV

Exclusion Criteria:

* Prior orthopedic surgery on the lower extremity or the trunk (<6 months)
* Prior neurosurgical interventions (<6 months)
* Significant mental retardation
* Severe contractures
* Prior Lokomat training (<6 months)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10-05 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
GMFM-66, section E | week 0, week 6, week 12

SECONDARY OUTCOMES:
GMFM-66, section D | week 0, week 6, week 12
Gait speed | week 0, week 6, week 12
6-minute walk test | week 0, week 6, week 12
3D gait analysis | week 0, week 6

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Ammann-Reiffer, MPTSc, Principal Investigator — University Children's Hospital Zurich, Rehabilitation Center Affoltern
Locations (2):
- Switzerland (2):
  - Paediatric Therapy Center Reha Rheinfelden, Rheinfelden, Canton of Aargau
  - University Children's Hospital Zurich, Rehabilitation Centre Affoltern, Affoltern am Albis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ammann-Reiffer C, Bastiaenen CHG, Meyer-Heim AD, van Hedel HJA. Lessons learned from conducting a pragmatic, randomized, crossover trial on robot-assisted gait training in children with cerebral palsy (PeLoGAIT). J Pediatr Rehabil Med. 2020;13(2):137-148. doi: 10.3233/PRM-190614. PMID 32444573
- [Derived] Ammann-Reiffer C, Bastiaenen CH, Meyer-Heim AD, van Hedel HJ. Effectiveness of robot-assisted gait training in children with cerebral palsy: a bicenter, pragmatic, randomized, cross-over trial (PeLoGAIT). BMC Pediatr. 2017 Mar 2;17(1):64. doi: 10.1186/s12887-017-0815-y. PMID 28253887